CLINICAL TRIAL: NCT07072104
Title: Longitudinal Assessment of Multidomain Reading-FREE Neurocognitive Markers for Early Detection of Developmental Dyslexia (FREE-DD)
Brief Title: Reading-FREE Markers for Early Detection of Developmental Dyslexia
Acronym: FREE-DD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: University of Urbino "Carlo Bo" (Other); University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Andrea Falini, Full Professor of Neuroradiology, Università Vita-Salute San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CET 501-2024; PRIN - Prot. 2022TA92HS (Other Grant/Funding Number: Ministry of University and Research - Projects of Significant National Interest (PRIN))
Record Dates: First submitted 2025-06-25; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Preterm Birth; Developmental Dyslexia
Keywords: Preterm birth; developmental dyslexia; reading-FREE; MRI; neurodevelopment
MeSH Terms: conditions — Premature Birth; Dyslexia

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment interventional model, involving two distinct groups: preterm-born (PTB) and term-born (ATB) children. Although no therapeutic intervention is administered, both groups undergo the same structured assessments at two time points, including behavioral screening, neuropsychological testing, and neuroimaging in Grade 2 and neuropsychological testing in Grade 3. The parallel design enables between-group comparisons to identify early neurocognitive and connectomic markers associated with the development of reading skills in children born preterm. The model supports hypothesis-driven evaluation of group-specific developmental trajectories using standardized procedures across cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTB (Experimental): Preterm-born children group
  Interventions: Behavioral: Multidomain Neuropsychological and Reading-Free Screening Tool (RSFT) Assessment Battery - Grade 2; Diagnostic Test: MRI - Grade 2; Behavioral: Multidomain Neuropsychological and Reading-Free Screening Tool (RSFT) Assessment Battery - Grade 3
- ATB (Experimental): At-term-born children group
  Interventions: Behavioral: Multidomain Neuropsychological and Reading-Free Screening Tool (RSFT) Assessment Battery - Grade 2; Diagnostic Test: MRI - Grade 2; Behavioral: Multidomain Neuropsychological and Reading-Free Screening Tool (RSFT) Assessment Battery - Grade 3

INTERVENTIONS:
Behavioral: Multidomain Neuropsychological and Reading-Free Screening Tool (RSFT) Assessment Battery - Grade 2 — * Behavioral testing: standardized neuropsychological battery (language, reading, attention, memory, intelligence)
  * RFST: Reading-Free Screening Tool assessing pre-reading cognitive markers
Diagnostic Test: MRI - Grade 2 — ■ Diagnostic Imaging: structural and resting-state functional MRI (T1-weighted and rs-fMRI)
Behavioral: Multidomain Neuropsychological and Reading-Free Screening Tool (RSFT) Assessment Battery - Grade 3 — * Behavioral testing: standardized neuropsychological battery (language, reading, attention, memory, intelligence)
  * RFST: Reading-Free Screening Tool assessing pre-reading cognitive markers

SUMMARY:
This study aims to identify early signs of developmental dyslexia (DD) and other reading difficulties in children born preterm, using behavioral, cognitive, and brain imaging data collected before reading problems typically become noticeable. Children born very early often face greater risk for reading and learning challenges, but these difficulties are not always detected in time for early support. This research seeks to fill that gap. A group of 30 children born preterm will be followed over time, alongside a control group of 15 children born at term. All children will be assessed during the second and third years of primary school (around ages 6-9). In Grade 2, children will undergo (a) a specially designed digital screening tool for reading difficulties that does not require actual reading (called the RFST), (b) standard tests of reading, language, and attention, and (c) structural and functional brain scans using Magnetic Resonance Imaging (MRI). In Grade 3, the children will be reassessed using the RFST and the cognitive and language tests. The goal is to identify specific behavioral and brain-based markers-particularly patterns of brain connectivity-that are already present in Grade 2 and can predict which children will go on to show reading difficulties in Grade 3. By comparing data from preterm and term-born children, researchers aim to discover early warning signs that are specific to children born preterm. By detecting these risks early, before reading delays become severe, the study hopes to guide new tools for screening and early intervention, tailored specifically to the unique developmental paths of children born preterm. This could help prevent later academic struggles and promote better long-term outcomes.

DETAILED DESCRIPTION:
This longitudinal study, titled "Longitudinal assessment of multidomain reading-FREE neurocognitive markers for early detection of Developmental Dyslexia (FREE-DD)", investigates early neurocognitive predictors of developmental dyslexia (DD) and related reading disorders in children born preterm (PTB), as compared to children born at term (ATB). Children born preterm are at elevated risk for neurodevelopmental vulnerabilities, including difficulties with language, attention, and reading acquisition, yet early identification of these risks remains limited.

The main objective of the study is to identify early connectomic and neurocognitive markers-obtained during second grade-that can predict the development of reading difficulties in PTB children by third grade. Particular emphasis is placed on connectomic features derived from functional and structural brain imaging, as well as on a specially designed behavioral tool: the Reading-Free Screening Tool (RFST), which assesses reading-related cognitive abilities without requiring the child to read.

The study adopts a prospective, longitudinal, monocentric cohort design, with two assessment waves:

* Grade 2 (Baseline/Timepoint 1): All enrolled children will undergo a comprehensive neuropsychological battery, RFST administration, and MRI acquisition (including structural and resting-state functional MRI).
* Grade 3 (Follow-up/Timepoint 2): Children will be reassessed using the RFST and neuropsychological tests to track changes in cognitive and reading-related abilities.

The study population includes 30 preterm-born (PTB) children and 15 term-born (ATB) children, all aged between 6 and 9 years, native Italian speakers, and right-handed. Children with structural brain lesions, congenital anomalies, or known neurological/psychiatric conditions will be excluded.

Primary Objective The primary goal is to determine whether functional brain network characteristics (measured via resting-state fMRI), along with morpho-structural, microstructural, and cognitive metrics collected at grade 2, can predict changes in RFST performance and reading skills between grade 2 and grade 3.

Secondary Objectives

Secondary aims include:

* Assessing correlations between functional connectivity and RFST indices.
* Evaluating whether measures of brain network segregation and integration can classify PTB vs. ATB readers and forecast individual developmental trajectories.
* Identifying multimodal predictors of atypical reading profiles across both grades.

Exploratory Objectives The study also seeks to explore the role of combined behavioral and neuroimaging data in outlining early neurocognitive trajectories specific to prematurity, which may indicate susceptibility to developmental dyslexia and related disorders. These exploratory outcomes will help refine developmental models and screening strategies.

Methodology

Participants will complete:

* Parental questionnaires (screening and developmental history),
* Manual preference testing,
* Two waves of neuropsychological assessments targeting language, attention, memory, phonological processing, and non-verbal intelligence,
* RFST administration,
* MRI scanning (T1-weighted structural imaging and resting-state fMRI). Data Analysis

Analysis will proceed in three main steps:

1. Functional Connectivity Mapping: Correlating ROI-to-ROI functional brain connectivity with RFST indices across all participants.
2. Group Classification: Extracting graph-based network metrics (e.g., segregation, integration) to classify PTB vs. ATB participants.
3. Predictive Modeling (PTB group): Employing the most relevant imaging and behavioral features to predict changes in RFST performance between grades 2 and 3, modeling individual developmental outcomes.

Timeline and Duration

* Enrollment Period: 2 months
* Total Participant Commitment: Approx. 4 hours (2 hours per visit across two school years)
* Study Duration: 10-12 months (including follow-up) This study is sponsored by the Università Vita-Salute San Raffaele and funded by PRIN (Progetti di Ricerca di Rilevante Interesse Nazionale - Bando 2022, Prot. 2022TA92HS). It will be conducted at the clinical center of the Ospedale San Raffaele (OSR), under the direction of the U.O. of Neuroradiology.

The findings from this study aim to inform the development of screening tools and targeted early interventions for children born preterm, potentially reducing the long-term impact of developmental dyslexia and enhancing academic and cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

For Preterm-Born (PTB) Children:

* Born preterm (i.e., gestational age < 39 weeks)
* Aged between 6 and 9 years at enrollment
* Absence of structural brain lesions (as assessed by prior clinical imaging)
* Italian as the first language (L1)
* Right-hand dominant
* Male or female

For At-Term-Born (ATB) Children:

* Born at term (i.e., gestational age between 39 and 42 weeks)
* Aged between 6 and 9 years at enrollment
* Absence of structural brain lesions (as assessed by prior clinical imaging)
* Italian as the first language (L1)
* Right-hand dominant
* Male or female

Exclusion Criteria:

For Preterm-Born (PTB) Children:

* History of congenital infections
* Diagnosis of Multiple Congenital Anomalies Syndrome
* Presence of focal intracerebral parenchymal lesions
* Pathological findings on conventional MRI

For At-Term-Born (ATB) Children:

* Presence of first-degree relatives diagnosed with developmental dyslexia (DD)
* Diagnosis of other learning or behavioral disorders
* Contraindications to MRI (e.g., metal implants, severe claustrophobia)

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in RFST Auditory Modality Composite Score From Grade 2 to Grade 3 in Preterm Children | From Grade 2 baseline to Grade 3 follow-up assessment (approx. 8-10 months)
  Composite score summarizing auditory-based sensorimotor, timing, discrimination, and inhibitory control abilities measured via the ReadFree Screening Tool (RFST) auditory modality tasks. Includes:
  * Auditory Reaction Time (median RTs of 8 trials)
  * Tapping and Entrainment to Metronome (tapping onset)
  * Free Tapping (motor rhythm without auditory cue)
  * Tone Discrimination (smallest perceptible pitch interval)
  * Cocktail Party Task (d-prime, target detection in multitalker noise)
  * Auditory Go/No-Go (d-prime, inhibition)
  * Auditory Anticipatory Timing (tapping onset accuracy) Each task is z-scored and aggregated into a single composite. Higher scores indicate better auditory sensorimotor and temporal processing.
Change in RFST Visual Modality Composite Score From Grade 2 to Grade 3 in Preterm Children | From Grade 2 baseline to Grade 3 follow-up assessment (approx. 8-10 months)
  Composite score summarizing visual-based sensorimotor, discrimination, and inhibitory control abilities from the RFST visual modality tasks. Includes:
  * Visual Reaction Time (median RTs of 8 trials)
  * Tapping and Entrainment to Visual Cue (tapping onset)
  * Free Tapping (motor rhythm without visual cue)
  * Grey-Scale Discrimination (smallest perceptible luminance interval)
  * Visual Go/No-Go (d-prime, visual inhibition)
  * Visual Anticipatory Timing (accuracy of tapping onset)
  * RAN-Shapes (number of shapes named in 30s) Each score is converted to z-units and averaged to yield a composite metric. Higher scores indicate better visual-motor and perceptual timing performance.
Grade 2 Composite Language Score in Preterm Children | Grade 2 baseline assessment
  A standardized composite language score derived from z-transformed or scalar scores of the following assessments:
  * Phoneme Deletion
  * BVL Auditory Discrimination (HIT-False Alarm Index, range: -100% to +100%)
  * NEPSY-II Subtests: L1, L3, L4, L5. The composite reflects mean z-scores (normalized against internal sample distribution) across all measures. Higher scores indicate better language functioning.
Grade 2 Composite Attention Score in Preterm Children | Grade 2 baseline assessment
  A composite attention score computed from standardized or scalar scores across the following assessments:
  * Colored Raven Matrices (Percentiles by age: 3rd-95th)
  * NEPSY-II Subtests:
    * A1 Visual Search
    * A2 Figural Fluency
    * A3 Auditory Attention
    * A4 Inhibition (Time; Accuracy)
    * A6 Categorization Each test is converted to a z-score and averaged for a domain-wide summary score. Higher scores indicate better attention performance.
Grade 2 Composite Reading Score in Preterm Children | Grade 2 baseline assessment
  Composite score combining metrics from multiple timed and accuracy-based reading assessments:
  * Lapel Reading Song (Words per minute: 21-157; Errors: 0-10)
  * PIN Reading (Words and Pseudo-words):
    * Reading Time
    * Syllables/sec
    * Number of Errors Each metric is z-normalized and averaged per task, then aggregated for a domain-level composite. Higher composite scores indicate better learning performance.
Grade 2 Resting-State fMRI Network Segregation Score in Preterm Children | Grade 2 baseline MRI session
  Resting-state functional connectivity-based modularity score, measuring the extent to which functional networks in the brain are subdivided into non-overlapping, highly interconnected communities. Higher modularity indicates greater network segregation.
Grade 2 Resting-State fMRI Network Integration Score in Preterm Children | Grade 2 baseline MRI session
  Participation coefficient derived from resting-state fMRI data, quantifying the extent to which brain nodes form diverse intermodular connections. Higher participation coefficient reflects greater network integration and communication between functional modules.

SECONDARY OUTCOMES:
Language Score at Grade 3 in Preterm Children | Grade 3 follow-up assessment
  The Peabody Picture Vocabulary Test (Italian version) is administered to assess receptive vocabulary. Raw scores are calculated by subtracting errors from the ceiling value. Age-standardized scores are derived from the raw score based on national norms. This outcome reflects language comprehension ability at Grade 3.
Composite Attention Score at Grade 3 in Preterm Children | Grade 3 follow-up assessment (8-10 months post-baseline)
  This outcome reflects attentional functioning based on multiple neuropsychological measures, aggregated as a domain-level composite. Tests include:
  * Mea Figural Fluency (percentiles)
  * Mea Cancellation (Sheets 5 & 10) (percentiles)
  * Mea PASOT (percentiles)
  * Mea Categorization (percentiles)
  * Colored Raven Matrices (age-based percentiles)
  * BVN Forward and Backward Span (z-scores or percentiles by age)
  * Prose Memory (number of correctly recalled morphological units; max 34)
  * VAUMELF - Repetition of Non-Words (correctness score, range: 0-40) Each test score is standardized (z-transformed or percentile-normalized as appropriate) and averaged into a single composite score representing domain-level attentional performance. Higher composite values indicate better attention function.
Composite Reading Score at Grade 3 in Preterm Children | Grade 3 follow-up assessment
  This outcome reflects reading and learning-related cognitive performance based on the following assessments:
  * MT3 Clinics Song Reading (Syllables/sec; number of errors; percentiles from 5th-90th)
  * DDE-2 Reading Words (z-score of speed and accuracy)
  * DDE-2 Reading Non-Words (z-scores of speed and accuracy)
  * BVSCO-3 Sentence Dictation (total errors; percentiles from 5th-95th)
  * AC-MT Judgment of Magnitude (number of correct responses; 5th-90th percentiles)
  * BDE-2 Triplets (total correct responses; clinical bands and percentile ranks)
  Each raw test score is converted to a standardized value (z-score or percentile), and the resulting values are averaged to produce a single composite score. Higher scores indicate better learning and reading competence.

OTHER OUTCOMES:
Grade 2 Global Efficiency Score from Resting-State Functional Connectivity in Preterm Children | Grade 2 baseline assessment
  Global efficiency is computed as the average inverse shortest path length across the entire resting-state functional connectivity network. It reflects the brain's capacity for parallel information transfer across distributed regions. Higher scores indicate greater global integration and reduced communication cost across brain regions.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Falini, Doctor of Medicine, Principal Investigator — 1. Vita-Salute San Raffaele University, Milan, Italy 2. Neuroradiology Unit and CERMAC, IRCCS Ospedale San Raffaele, Milan, Italy
Locations (1):
- Neuroradiology Unit and CERMAC, IRCCS Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canini, M., Cara, C., Oprandi, C., Katušić, A., Žunić Išasegi, I., Messina, A., Zambon, A. A., Pecco, N., Barni, S., Poloniato, A., Natali Sora, M. G., Falautano, M., Scifo, P., Barera, G., Tettamanti, M., Falini, A., Baldoli, C., & Della Rosa, P. A. (2025). Functional connectivity markers of prematurity at birth predict neurodevelopmental outcomes at 6, 12, 24, and 36 months. International Journal of Behavioral Development, 0(0). https://doi.org/10.1177/01650254241312136
- [Background] Della Rosa PA, Canini M, Marchetta E, Cirillo S, Pontesilli S, Scotti R, Natali Sora MG, Poloniato A, Barera G, Falini A, Scifo P, Baldoli C. The effects of the functional interplay between the Default Mode and Executive Control Resting State Networks on cognitive outcome in preterm born infants at 6 months of age. Brain Cogn. 2021 Feb;147:105669. doi: 10.1016/j.bandc.2020.105669. Epub 2020 Dec 17. PMID 33341657
- [Background] Baldoli C, Scola E, Della Rosa PA, Pontesilli S, Longaretti R, Poloniato A, Scotti R, Blasi V, Cirillo S, Iadanza A, Rovelli R, Barera G, Scifo P. Maturation of preterm newborn brains: a fMRI-DTI study of auditory processing of linguistic stimuli and white matter development. Brain Struct Funct. 2015 Nov;220(6):3733-51. doi: 10.1007/s00429-014-0887-5. Epub 2014 Sep 23. PMID 25244942
- [Background] Carioti D, Stucchi NA, Toneatto C, Masia MF, Del Monte M, Stefanelli S, Travellini S, Marcelli A, Tettamanti M, Vernice M, Guasti MT, Berlingeri M. The ReadFree tool for the identification of poor readers: a validation study based on a machine learning approach in monolingual and minority-language children. Ann Dyslexia. 2023 Oct;73(3):356-392. doi: 10.1007/s11881-023-00287-3. Epub 2023 Aug 7. PMID 37548832